CLINICAL TRIAL: NCT03816631
Title: A Phase 1, Open-label, Single-dose Study to Evaluate the Effect of Hepatic Impairment on the Pharmacokinetics of Orally Administered Pimodivir in Adult Subjects
Brief Title: A Study of Orally Administered Pimodivir in Adult Participants With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108571; 2018-002817-36 (EudraCT Number); 63623872FLZ1013 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — pimodivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: Group 1: Severe hepatic function (Experimental): Participants with severe hepatic function will receive single oral dose of pimodivir 600 milligram (mg) (2*300 mg tablet) under fasted condition on Day 1.
  Interventions: Drug: Pimodivir
- Part A and B: Group 2: Normal hepatic function (Experimental): Participants with normal hepatic function will receive single oral dose of pimodivir 600 mg (2*300 mg tablet) under fasted condition on Day 1. The recruitment in Part B will be started based on assessment by Sponsor upon evaluation of partial data obtained in Part A.
  Interventions: Drug: Pimodivir
- Part B: Group 3: Moderate hepatic function (Experimental): Participants with moderate hepatic function will receive single oral dose of pimodivir 600 mg (2*300 mg tablet) under fasted condition on Day 1. The recruitment in Part B will be started based on assessment by Sponsor upon evaluation of partial data obtained in Part A.
  Interventions: Drug: Pimodivir
- Part B: Group 4: Mild hepatic function (Experimental): Participants with mild hepatic function will receive single oral dose of Pimodivir 600 mg (2*300 mg tablet) under fasted condition on Day 1. The recruitment in Part B will be started based on assessment by Sponsor upon evaluation of partial data obtained in Part A.
  Interventions: Drug: Pimodivir

INTERVENTIONS:
Drug: Pimodivir — Participants will receive single oral dose of Pimodivir 600 mg (2*300 mg tablets) under fasted condition on Day 1.
  Other Names: JNJ-63623872

SUMMARY:
The purpose is to evaluate the pharmacokinetics (PK) of a single oral dose of 600 milligram (mg) pimodivir in adult participants with impaired hepatic function compared to adult participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a stable hepatic function as confirmed by albumin levels, prothrombin time (PT), International Normalized Ratio (INR), and platelet count measured during screening and those measured within 24 hours prior to study drug administration. Participants with a Transjugular Intrahepatic Portosystemic Shunt procedure will be allowed to participate in the study
* Participant must have a body mass index (BMI; weight [Kilogram {kg}/height^2 [meter {m}^2]) between 18.0 and 38.0 kg/m^2, extremes included, and body weight not less than 50 kg at screening
* Participant must have a 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function at screening, including: (a) Sinus rhythm; (b) Pulse rate between 45 and 100 beats per minute (bpm); (c) QT interval corrected for heart rate (QTc) according to Fridericia formula (QTcF) less than or equal to (<=) 450 millisecond (ms) for male participant and <= 470 ms for female participant; (d) QRS interval of less than (<) 120 ms; (e) PR interval <= 220 ms and (f) Electrocardiogram morphology consistent with healthy cardiac conduction and function. Participant with pacemaker is eligible as long as all criteria mentioned above are met
* A woman, except if postmenopausal, must have a negative highly sensitive serum pregnancy test (beta-human chorionic gonadotropin [beta-hCG]) at screening and a negative urine pregnancy test on Day -1
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies

Exclusion Criteria:

* Participant has known allergies, hypersensitivity, or intolerance to pimodivir or its excipients
* Participant has donated blood or blood products or had substantial loss of blood (more than 500 milliliter [mL]) within 3 months before administration of the study drug or intention to donate blood or blood products during the study
* Participant has received an experimental drug (including investigational vaccines) or used an experimental medical device within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before administration of the study drug is scheduled
* Participant has preplanned surgery or procedures that would interfere with the conduct of the study
* Participant is a woman who is pregnant, breast-feeding, or planning to become pregnant while enrolled in this study or a woman of childbearing potential who is unwilling to use an acceptable method of contraception

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration (Cmax) of Pimodivir | Predose, 30 min, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96, 120 hours post dose and end of study (up to Day 14)
  Cmax is defined as maximum observed analyte concentration of pimodivir.
Area Under Concentration-Time Curve from Time 0 to the Time of the Last Concentration (AUC[last]) of Pimodivir | Predose, 30 min, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96, 120 hours post dose and end of study (up to Day 14)
  AUC(last) is defined as the time 0 to the time of the last measurable (non-below quantification limit) concentration of Pimodivir calculated by linear-linear trapezoidal summation.
Area Under Concentration-Time Curve from Time 0 to Infinite Time (AUC[0-infinity]) of Pimodivir | Predose, 30 min, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72, 96, 120 hours post dose and end of study (up to Day 14)
  The AUC ([0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C (last)/ lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to the time of the last measurable concentration, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants with Adverse Event as a Measure of Safety and Tolerability | Approximately 42 days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (2):
- Germany (2):
  - CRS Clinical Research Services Kiel GmbH, Kiel
  - APEX GmbH, München

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency